CLINICAL TRIAL: NCT00377260
Title: Efficacy of Antimicrobials in Young Children With Acute Otitis Media (AOM)
Brief Title: Acute Otitis Media (AOM) Therapy Trial in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Alejandro Hoberman, Chief, Division of General Academic Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-0142; U01AI066007 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Acute Otitis Media
Keywords: acute otitis media, infants, children
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin-clavulanate (Experimental): Reconstituted amoxicillin-clavulanate at 90/6.4 mg/kg/day in 2 divided doses for 10 days.
  Interventions: Drug: amoxicillin-clavulanate
- Placebo (Placebo Comparator): Reconstituted placebo in 2 divided doses for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: amoxicillin-clavulanate — Augmentin ES-600™: Amoxicillin-clavulanate potassium (600/42.9 mg per 5 mL), administered at a dose of 90/6.4 mg/kg/day in 2 divided doses for 10 days with strawberry cream flavor.
  Other Names: Augmentin; amox-clav
  Arms: Amoxicillin-clavulanate
Drug: Placebo — Same base formulation of the licensed product Augmentin ES-600™, with the same strawberry cream flavor.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn whether or not all children with ear infections (acute otitis media or AOM) should be treated with antibiotics. The study will compare two treatment strategies, "watchful waiting" or treatment with antibiotics, to determine which is more appropriate for children with AOM. About 268 children in Pittsburgh, between the ages of 6-23 months, with AOM will be enrolled in the study. They will be treated either with Augmentin (an antibiotic) or placebo for 10 days and closely followed for about 1 month. Parents will be asked to write information about their child in a Patient Diary. A general physical exam, including an ear exam, will be performed 4 times during the study. A mucus sample will be collected from the back of each child's nose. Parents will be asked questions during phone calls and at every visit. If a child has not improved or has worsened, the investigators will prescribe a different antibiotic that is known to kill resistant germs.

DETAILED DESCRIPTION:
The purpose of this randomized, double-masked, placebo-controlled, single-center clinical trial is to determine the efficacy of antimicrobials in young children with acute otitis media (AOM). The primary objectives are to compare time to resolution of symptoms (initial and sustained) in children receiving amoxicillin-clavulanate (90/6.4mg/kg/day in 2 divided doses for 10 days) to children receiving placebo (in 2 divided doses for 10 days), and to compare the weighted average AOM-Severity of Symptoms (AOM-SOS) scores in the two groups during days 1-7. The secondary objectives are to: evaluate the clinical efficacy of amoxicillin-clavulanate vs. placebo at the on-therapy visit (Day 4-5, and at least 72 hours after initial dose of study medication); evaluate the clinical efficacy of amoxicillin-clavulanate vs. placebo at the end-of-therapy visit (Day 10-12); compare AOM-SOS and AOM-Faces scales between treatment groups during each of the first 7 days of therapy and at all study visits; compare the proportion of children in each treatment group who develop worsening symptoms before having received 72 hours of study medication; compare the two treatment groups regarding the quantity of analgesic medication administered by children's parents; compare the incidence of adverse events accompanying the two treatment regimens; compare the effects of amoxicillin-clavulanate vs. placebo on the overall proportion of children with nasopharyngeal (NP) colonization with AOM pathogens (S. pneumoniae, H. influenzae, M. catarrhalis, S. pyogenes), and on the proportion of children with NP colonization with penicillin non-susceptible S. pneumoniae; compare the 2 treatment groups regarding tympanometric outcomes at the on-therapy (Day 4-5), end-of-therapy (Day 10-12) and follow-up (Day 21-25) visits, using an algorithm that permits estimation of the probability of middle ear effusion given any particular tympanographic configuration; compare direct and indirect medical costs between the two treatment groups; and compare parental satisfaction with therapy between the two treatment groups. Participants will include 268 children, aged 6 to 23 months, diagnosed with acute otitis media in Western Pennsylvania. These participants will be recruited into the study at Children's Hospital of Pittsburgh (CHP), Pittsburgh, PA, and Armstrong Pediatrics (Children's Community Pediatrics: an affiliate of CHP) in Kittanning, PA. Subjects will be randomized to receive either amoxicillin-clavulanate or placebo twice daily for 10 days. Parents of the subject will be asked to track symptom status, medication use (study medication and acetaminophen), fever and diarrhea in a study memory aid. Study procedures will include a medical history, vital signs, weight, clinical information regarding signs and symptoms of infection, nasopharyngeal specimens, and a physical exam including tympanometry. Each child will be examined three additional times: 4-5 days after starting the medicine, study day 10-12 and 21-25 days after enrolling in the study. During these visits, study staff will review the child's symptoms and examine the child's ears. The study staff will also obtain a nasopharyngeal culture in order to look for resistant bacteria and to make appropriate changes in antibiotic treatment. Daily telephone assessments will be made by study staff on days 2, 3, and 4 of therapy to make sure the child is getting better. The study staff will see a child anytime a parent feels their child has not improved or has worsened.

ELIGIBILITY:
Inclusion Criteria:

* aged 6 to 23 months
* have received at least two doses of pneumococcal conjugate vaccine (Prevnar) and Haemophilus influenzae type B vaccine
* have evidence of acute otitis media (AOM) defined as:

  1. Recent (within 48 hours), onset of signs and symptoms and a score of greater than or equal to 3 on the AOM-SOS scale.
  2. Middle ear effusion evidenced by at least two of the following:
* decreased or absent tympanic membrane mobility by pneumatic otoscopy,
* yellow or white discoloration of the tympanic membrane,
* opacification of the tympanic membrane, plus
* 1+ bulging of the tympanic membrane with either marked erythema or otalgia, or
* 2+ or 3+ bulging of the tympanic membrane

Exclusion Criteria:

* certain signs or symptoms (e.g., toxic appearance [capillary refill greater than 3 seconds, systolic blood pressure less than 60 mm Hg], otalgia for a period greater than 48 hours, spontaneous perforation of the tympanic membrane and drainage or temperature greater than or equal to 105 degrees F);
* clinical or anatomical characteristics that might obscure response to treatment (e.g., tympanostomy tube[s] in place or a history of tympanostomy tubes, unrepaired or repaired overt or submucous cleft palate, high-arched palate, or Down's syndrome);
* underlying systemic problems that might obscure response to infection (e.g., serious underlying disease [e.g., cystic fibrosis, neoplasm, juvenile diabetes]), concomitant infection that would preclude evaluation of the response of the child's AOM to study medication, known renal insufficiency (i.e., serum creatinine greater than or equal to 1.5 times upper limit of normal for age), known hepatic insufficiency or a history of amoxicillin-clavulanate-associated cholestatic jaundice or hepatic dysfunction, history of immune dysfunction, deficiency or receipt of immunosuppressive therapy, chronic gastrointestinal conditions (i.e., malabsorption, inflammatory bowel disease), malignancy;
* sensorineural hearing loss either unilateral or bilateral;
* comedications (e.g., systemic corticosteroids at any point while enrolled in the study, more than one dose of systemic antimicrobial therapy within 96, any investigational drug or vaccine;
* hypersensitivity to penicillin, amoxicillin or amoxicillin-clavulanate, or phenylketonuria or known hypersensitivity to aspartame;
* unable to complete the study protocol or not having access to a telephone; and
* current enrollment in another study or previously enrolled in this study.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 291 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Hoberman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaikh N, Hoberman A, Paradise JL, Rockette HE, Kurs-Lasky M, Martin JM. Association Between Nasopharyngeal Colonization and Clinical Outcome in Children With Acute Otitis Media. Pediatr Infect Dis J. 2023 Aug 1;42(8):e274-e277. doi: 10.1097/INF.0000000000003956. Epub 2023 Apr 26. PMID 37171965
- [Derived] Hoberman A, Paradise JL, Rockette HE, Shaikh N, Wald ER, Kearney DH, Colborn DK, Kurs-Lasky M, Bhatnagar S, Haralam MA, Zoffel LM, Jenkins C, Pope MA, Balentine TL, Barbadora KA. Treatment of acute otitis media in children under 2 years of age. N Engl J Med. 2011 Jan 13;364(2):105-15. doi: 10.1056/NEJMoa0912254. PMID 21226576
- [Derived] Hoberman A, Paradise JL, Shaikh N, Greenberg DP, Kearney DH, Colborn DK, Rockette HE, Kurs-Lasky M, McEllistrem MC, Zoffel LM, Balentine TL, Barbadora KA, Wald ER. Pneumococcal resistance and serotype 19A in Pittsburgh-area children with acute otitis media before and after introduction of 7-valent pneumococcal polysaccharide vaccine. Clin Pediatr (Phila). 2011 Feb;50(2):114-20. doi: 10.1177/0009922810384259. Epub 2010 Nov 22. PMID 21098526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited over 3 respiratory seasons, beginning on 11/31/2006 with the last enrollment on 3/31/2009. There were 2 enrollment sites, as well as referrals from private pediatricians. One site was a large private practice; the other was a large hospital based practice. This was for generalizability.
Pre-assignment Details: There were 2 children who signed consents but were not randomized. One parent withdrew consent and one child, referred from an outside practice, was found to not be eligible.
Period: Overall Study
Arm/Group | Amoxicillin-Clavulanate | Placebo
Started | 144 | 147
Completed | 142 (A child is considered a completer if he/she had at least one visit after the end of therapy.) | 142 (A child is considered a completer if he/she had at least one visit after the end of therapy.)
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin-Clavulanate | Placebo | Total
Number analyzed (Participants) | 144 | 147 | 291
Age, Customized [Number; unit: participants]
  6-11 months | 83 | 78 | 161
  12-17 months | 35 | 42 | 77
  18-23 months | 26 | 27 | 53
Gender [Count of Participants; unit: Participants]
  Female | 69 | 67 | 136
  Male | 75 | 80 | 155
Colonization With AOM Pathogens [Number; unit: participants] — AOM pathogens refer to Streptococcus Pneumoniae, Haemophilus Influenzae, Moraxella Catarrhalis or Streptococcus Pyogenes
  participants
    Presence of at least one AOM pathogen | 123 | 119 | 242
    Absence of any AOM pathogen | 16 | 24 | 40
    No culture result | 5 | 4 | 9
Degree of tympanic membrane bulging [Number; unit: participants] — The degree of bulging for the ear with the greater level of bulging at entry is summarized. The otoscopists rated this as slight bulging, moderate bulging or marked bulging. The otoscopists have all been validated for inter-observer reliability.
  participants
    Slight | 42 | 39 | 81
    Moderate | 63 | 70 | 133
    Marked | 39 | 38 | 77
Ethnicity [Number; unit: participants] — Parents were asked if their child is Hispanic.
  participants
    Hispanic | 21 | 19 | 40
    Non-Hispanic | 123 | 128 | 251
Exposed to other children [Number; unit: participants] — Exposed to other children is defined as a child being exposed to 3 or more children, including siblings, for at least 10 hours per week.
  Not exposed is defined as any child who does not meet this criteria.
  participants
    Exposed | 69 | 72 | 141
    Not exposed | 75 | 75 | 150
Health insurance status [Number; unit: participants] — Parents were asked the child's health insurance status
  participants
    Private | 43 | 42 | 85
    Medicaid | 98 | 103 | 201
    None | 3 | 2 | 5
History of recurrent acute otitis media [Number; unit: participants] — Records were obtained and reviewed for a history of recurrent acute otitis media.
  "Yes" indicates that the child had a documented history of at least 3 acute otitis media episodes in the past 6 months or at least 4 episodes in the past year.
  "No" indicates that the child did not meet the criteria for "Yes".
  participants
    Yes | 21 | 29 | 50
    No | 123 | 118 | 241
Laterality of Acute Otitis Media [Number; unit: participants] — Bilateral means that both ears were found to be acute. Unilateral means that only one ear was found to be acute, the other ear could have had middle ear effusion or have been free of middle ear effusion.
  participants
    Bilateral | 75 | 77 | 152
    Unilateral | 69 | 70 | 139
Maternal Education [Number; unit: participants] — Parents were asked about the highest level of maternal education.
  participants
    Less than high school | 24 | 16 | 40
    High school graduate | 90 | 95 | 185
    College graduate | 30 | 35 | 65
    Unknown | 0 | 1 | 1
Race [Number; unit: participants] — Parents were asked what race or races they would use to describe their child. Caucasian and African-American are listed when only one race was given. Other includes other races as well as any who gave more than one race.
  participants
    Caucasian | 66 | 65 | 131
    African-American | 62 | 58 | 120
    Other | 16 | 24 | 40
Severity of symptoms score [Number; unit: participants] — Parents completed the Acute Otitis-Media-Severity of Symptoms (AOM-SOS)scale prior to their child's ear exam. It's a list of 7 symptoms associated with Acute Otitis-media.
  [tugging/rubbing/holding ears; crying more; irritable/fussy; difficulty sleeping; less playful/active; eating less; fever or warm to touch. The parent rates these symptoms as No (0 points), A little (1 point) or A lot (2 points). Children must have at least 3 points to qualify, so the minimum score is 3, the maximum is 14.
  participants
    Score of 3-5 | 37 | 33 | 70
    Score of 6-8 | 46 | 51 | 97
    Score of 9-11 | 46 | 44 | 90
    Score of 12-14 | 15 | 19 | 34
Study Site [Number; unit: participants] — Children's Hospital of Pittsburgh (CHP) is the Primary Care Center of CHP. Armstrong Pediatrics is a large community practice in Kittanning, PA.
  participants
    Children's Hospital of Pittsburgh (Pittsburgh, PA) | 113 | 117 | 230
    Armstrong Pediatrics (Kittanning, PA) | 31 | 30 | 61
Mean Estimated Probability of Middle Ear Effusion [Mean (Standard Deviation); unit: probability of effusion] — For tympanograms with values for height, middle-ear air pressure, and gradient width, the probability of Middle Ear Effusion (MEE) was estimated by applying an algorithm developed by Smith et al. If the tympanogram was flat and had no printed values for the 3 fields, the probability of MEE was estimated to be .802 based on the proportion of ears with flat graphs that were found otoscopically, by Smith et al, to have MEE.
  probability of effusion
    Right ear | .42 (.31) | .39 (.27) | .41 (.29)
    Left ear | .35 (.30) | .44 (.29) | .40 (.30)
Mean score of AOM-SOS [Mean (Standard Deviation); unit: AOM-SOS score] — This is the mean score for each arm. Parents completed the Acute Otitis Media -Severity of Symptoms (AOM-SOS) scale prior to their child's ear exam. It's a list of 7 symptoms associated with Acute Otitis-media.
  [tugging/rubbing/holding ears; crying more; irritable/fussy; difficulty sleeping; less playful/active; eating less; fever or warm to touch. The parent rates these symptoms as No (0 points), A little (1 point) or A lot (2 points). Children must have at least 3 points to qualify, so the minimum score is 3, the maximum is 14.
  AOM-SOS score | 7.69 (2.85) | 7.90 (2.87) | 7.80 (2.86)

OUTCOME MEASURES:

1. Secondary Outcome: The Distribution of Clinical Failures by the On-therapy Visit According to Treatment Assignment
Description: Clinical failure by the on-therapy visit is defined as either failure to achieve substantial improvement in symptoms, or worsening of otoscopic signs, or both.
Time Frame: On-therapy visit. The mean day for this visit was 5.0.
Population: The analysis was ITT. The number of participants equals the number of children followed at least 72 hours after the initial dose of study medication plus the number of children meeting the criteria for clinical failure less than 72 hours after the initial dose of study medication.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 145
participants
  Clinical failures by the on therapy visit | 5 | 34
  Subjects not classified as clinical failures | 138 | 111
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of clinical treatment failures by the on-therapy visit; Test type: Superiority or Other; p < .001, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

2. Secondary Outcome: The Distribution of Clinical Failures by the End-of-therapy Visit According to Treatment Assignment
Description: Clinical failure by the end of therapy visit is defined as failure to achieve complete or virtually complete resolution of symptoms and of otoscopic signs, but without regard to the persistence of middle ear effusion.
Time Frame: End-of-therapy visit. The mean day for this visit was 11.6.
Population: The analysis was ITT. The number of participants equals the number of children evaluated post therapy plus the number of children who met the criteria for clinical failure prior to the end of therapy.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 142 | 143
participants
  Clinical failures by the end of therapy visit | 23 | 73
  Subjects not classified as clinical failures | 119 | 70
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of clinical failures by the end of therapy; Test type: Superiority or Other; p < .001, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

3. Secondary Outcome: The Mean Acute Otitis Media - Severity of Symptom (AOM-SOS) Score, Post-enrollment, Over the First 7 Days of Therapy According to Treatment Assignment
Description: The parent rated each of 7 symptoms (ear tugging, crying, irritability, difficulty sleeping, diminished activity, diminished appetite & fever) as 0, 1 or 2 (none, a little, a lot) and recorded the ratings in a diary following enrollment on Day 1, twice daily Days 2 and 3, then once daily Days 4-7. Each set of ratings was summed to obtain an AOM-SOS score as a measure of symptom burden. The maximum possible score was 14 and the minimum was 0.
Time Frame: During the first 7 days of therapy
Population: The analysis was ITT. The number of participants equals the number of children with at least one AOM-SOS score post-enrollment in the first 7 days of therapy. The score was based on AM and PM diaries completed at home by the child's parent.
Measure: Mean (Standard Deviation); unit: AOM-SOS score
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 144
AOM-SOS score
  Day 1 PM | 5.80 (3.61) | 6.20 (3.33)
  Day 2 AM | 4.12 (3.06) | 4.85 (3.54)
  Day 2 PM | 3.78 (3.05) | 4.33 (3.41)
  Day 3 AM | 2.86 (2.69) | 3.37 (3.04)
  Day 3 PM | 2.82 (2.67) | 3.25 (2.94)
  Day 4 | 2.40 (2.62) | 2.68 (2.59)
  Day 5 | 1.93 (2.09) | 2.41 (2.59)
  Day 6 | 1.40 (1.69) | 2.31 (2.29)
  Day 7 | 1.28 (1.64) | 1.94 (2.50)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the symptom burden as measured by the respective mean scores over time; Test type: Superiority or Other; p = .02, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

4. Secondary Outcome: The Distribution of Children Developing Worsening Symptoms Prior to Receiving 72 Hours of Study Medication According to Treatment Assignment
Description: The parent rated each of 7 symptoms (ear tugging, crying, irritability, difficulty sleeping, diminished activity, diminished appetite & fever) as 0, 1 or 2 (none, a little, a lot) and recorded the ratings in a diary following enrollment on Day 1 and twice daily Days 2 and 3. Each set of ratings was summed to obtain an Acute Otitis Media-Severity of Symptoms (AOM-SOS) score. We compared a child's AOM-SOS scores in the first 72 hours to his/her score at enrollment to determine if a child's symptoms got worse (score increased) or remained unchanged or improved (score remained same or decreased).
Time Frame: Before receiving 72 hours of study medication
Population: The analysis was ITT. The number of participants equals the number of children with follow-up whose parent(s) recorded AM and/or PM symptom scores in the first 3 days of treatment.
Measure: Number; unit: Participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 143
Participants
  Number of children with worsening symptoms | 31 | 39
  Number of children unchanged or improved | 112 | 104
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of children who develop worsening symptoms within the first 3 days of treatment; Test type: Superiority or Other; p = .24, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

5. Secondary Outcome: The Mean Number of Times Analgesic Medication Was Administered to the Child According to Treatment Assignment
Description: The parents were asked to complete a memory aid for the first 10 days of the study. One item asked them to record medications administered to the child in addition to the study medication. The data presented shows the mean number of times analgesic, i.e. ibuprofen or acetaminophen, was administered.
Time Frame: The first 10 days of follow-up
Population: The analysis was ITT. The participants for analysis were the children with follow-up.
Measure: Mean (Standard Deviation); unit: times analgesic was administered
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 146
times analgesic was administered | .37 (.48) | .43 (.48)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the average number of doses of analgesic medication administered by parents; Test type: Superiority or Other; p = .35, Regression, Linear — A weighted regression model was used with weights equal to the number of days information regarding analgesic use was reported by the parents; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

6. Secondary Outcome: The Distribution of Children With Observed or Parent Reported Adverse Events or Complications According to Treatment Assignment
Description: Analysis was limited to those adverse events identified as being associated with either the study medication or the antimicrobials administered to children who were treatment failures or as being a complication of acute otitis media.
Time Frame: We monitored children and queried parents regarding adverse events at each study visit, i.e. Day 4-5, Day 10-12, and Day 21-25, and at interim visits. The last assessment was made at the Day 21-25 visit. The mean day for this visit was 22.8.
Population: The analysis was ITT. The number of participants equals the number of children randomized.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 144 | 147
participants
  Mastoiditis | 0 | 1
  Perforation of tympanic membrane | 1 | 7
  Protocol-defined diarrhea | 36 | 22
  Diaper dermatitis | 73 | 51
  Oral thrush | 7 | 1
  Vomiting | 12 | 12
  Rash | 1 | 2
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with protocol-defined diarrhea; Test type: Superiority or Other; p = .04, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 2: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with diaper dermatitis; Test type: Superiority or Other; p < .01, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 3: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with oral thrush; Test type: Superiority or Other; p = .07, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 4: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with vomiting; Test type: Superiority or Other; p > .99, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 5: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with rash; Test type: Superiority or Other; p > .99, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 6: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with mastoiditis; Test type: Superiority or Other; p = .99, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 7: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the proportion of children with perforation of their tympanic membrane; Test type: Superiority or Other; p = .08, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

7. Secondary Outcome: The Distribution of Children With Nasopharyngeal (NP) Colonization With AOM Pathogens at the End-of-therapy Visit According to Treatment Assignment
Description: AOM pathogens are defined as Streptococcus Pneumoniae or Haemophilus Influenzae or Moraxella Catarrhalis or Streptococcus Pyogenes. Nasopharyngeal cultures were obtained at the end of therapy visit.
Time Frame: End-of-therapy visit. The mean day for this visit was 11.6.
Population: The analysis was ITT. The number of participants equals the number of children with NP culture results at the end-of-therapy visit.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 130 | 131
participants
  Presence of at least one AOM pathogen | 63 | 88
  Absence of any AOM pathogen | 67 | 43
  Presence of Streptococcus pneumoniae | 18 | 46
  Absence of Streptococcus pneumoniae | 112 | 85
  Presence of Haemophilus influenzae | 45 | 44
  Absence of Haemophilus influenzae | 85 | 87
  Presence of Moraxella catarrhalis | 9 | 38
  Absence of Moraxella catarrhalis | 121 | 93
  Presence of Streptococcus pyogenes | 0 | 3
  Absence of Streptococcus pyogenes | 130 | 128
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of culture results with at least one AOM pathogen present; Test type: Superiority or Other; p = .002, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 2: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of culture results with Streptococcus pneumoniae present; Test type: Superiority or Other; p < .001, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 3: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of culture results with Haemophilus influenzae present; Test type: Superiority or Other; p = .85, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 4: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of culture results with Moraxella catarrhalis present; Test type: Superiority or Other; p < .001, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 5: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of culture results with Streptococcus pyogenes present; Test type: Superiority or Other; p = .28, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

8. Secondary Outcome: The Distribution of Children With Nasopharyngeal (NP) Colonization With Penicillin-susceptible Streptococcus Pneumoniae (S. pn) at the End-of-therapy Visit According to Treatment Assignment
Time Frame: End-of-therapy visit. The mean day for this visit was 11.6.
Population: The analysis was ITT. The number of participants equals the number of children with NP culture results and results regarding penicillin susceptibility at the end-of-therapy visit.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 130 | 130
participants
  Colonization with penicillin-susceptible S. pn | 1 | 28
  No colonization with penicillin-susceptible S. pn | 129 | 102
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the proportion of children colonized with penicillin-susceptible Streptococcus pneumoniae; Test type: Superiority or Other; p < .001, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

9. Secondary Outcome: The Distribution of Children With Nasopharyngeal (NP) Colonization With AOM Pathogens at the Follow-up Visit According to Treatment Assignment
Description: AOM pathogens are defined as Streptococcus Pneumoniae or Haemophilus Influenzae or Moraxella Catarrhalis or Streptococcus Pyogenes. Nasopharyngeal cultures were obtained at the follow-up visit.
Time Frame: Follow-up visit. The mean day for this visit was 22.8.
Population: The analysis was ITT. The number of participants equals the number of children with NP culture results at the follow-up visit.
Measure: Number; unit: participant
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 128 | 130
participant
  Presence of at least one AOM pathogen | 76 | 89
  Absence of any AOM pathogen | 52 | 41
  Presence of Streptococcus pneumoniae | 26 | 42
  Absence of Streptococcus pneumoniae | 102 | 88
  Presence of Haemophilus influenzae | 38 | 38
  Absence of Haemophilus influenzae | 90 | 92
  Presence of Moraxella catarrhalis | 29 | 31
  Absence of Moraxella catarrhalis | 99 | 99
  Presence of Streptococcus pyogenes | 1 | 0
  Absence of Streptococcus pyogenes | 127 | 130
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = .10, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 2: Comparison: Amoxicillin-Clavulanate vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = .03, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 3: Comparison: Amoxicillin-Clavulanate vs Placebo; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p = .96, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 4: Comparison: Amoxicillin-Clavulanate vs Placebo; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = .79, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children
Statistical Analysis 5: Comparison: Amoxicillin-Clavulanate vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = .98, Regression, Logistic; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

10. Secondary Outcome: The Distribution of Children With Nasopharyngeal (NP) Colonization With Penicillin-susceptible Streptococcus Pneumoniae (S. pn) at the Follow-up Visit
Time Frame: Follow-up visit. The mean day for this visit was 22.8.
Population: The analysis was ITT. The number of participants equals the number of children with NP culture results and results regarding penicillin susceptibility at the follow-up visit.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 128 | 129
participants
  Colonization with penicillin-susceptible S. pn | 7 | 17
  No colonization with penicillin-susceptible S. pn | 121 | 112
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = .04, Regression, Logistic; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

11. Secondary Outcome: The Probability of Middle Ear Effusion, Based on an Algorithm That Estimates the Probability of Middle Ear Effusion From an Interpretable Tympanographic Configuration, at the On-therapy Visit According to Treatment Assignment
Description: For tympanograms with values for height, middle-ear air pressure, and gradient width, the probability of Middle Ear Effusion (MEE) was estimated by applying an algorithm developed by Smith et al. If the tympanogram was flat and had no printed values for the 3 fields, the probability of MEE was estimated to be .802 based on the proportion of ears with flat graphs that were found otoscopically, by Smith et al, to have MEE.
Time Frame: On-therapy visit. The mean day for this visit was 5.0.
Population: The analysis was ITT. The number of participants equals the number of children for which at least one ear has an interpretable tympanogram at the on-therapy visit.
Measure: Mean (Standard Deviation); unit: probability of effusion
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 121 | 121
probability of effusion
  Right ear | .36 (.29) | .42 (.29)
  Left ear | .39 (.31) | .48 (.29)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the probability of middle ear effusion at the on-therapy visit; Test type: Superiority or Other; p = .03, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

12. Secondary Outcome: The Probability of Middle Ear Effusion, Based on an Algorithm That Estimates the Probability of Middle Ear Effusion From an Interpretable Tympanographic Configuration, at the End-of-therapy Visit According to Treatment Assignment
Description: as for outcome 11
Time Frame: End-of-therapy visit. The mean day for this visit was 11.6.
Population: The analysis was ITT. The number of participants equals the number of children for which at least one ear has an interpretable tympanogram at the end-of-therapy visit.
Measure: Mean (Standard Deviation); unit: probability of effusion
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 120 | 119
probability of effusion
  Right ear | .32 (.27) | .41 (.28)
  Left ear | .33 (.28) | .41 (.27)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the probability of middle ear effusion at the end-of-therapy visit; Test type: Superiority or Other; p = .006, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

13. Secondary Outcome: The Probability of Middle Ear Effusion, Based on an Algorithm That Estimates the Probability of Middle Ear Effusion From an Interpretable Tympanographic Configuration, at the Follow-up Visit According to Treatment Assignment
Description: as for outcome 11
Time Frame: Follow-up visit. The mean day for this visit was 22.8.
Population: The analysis was ITT. The number of participants equals the number of children for which at least one ear has an interpretable tympanogram at the follow-up visit.
Measure: Mean (Standard Deviation); unit: probability of effusion
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 129 | 121
probability of effusion
  Right ear | .28 (.28) | .32 (.29)
  Left ear | .27 (.30) | .37 (.31)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; The analysis was ITT. The number of participants equals the number of children for which at least one ear has an interpretable tympanogram at the follow-up visit; Test type: Superiority or Other; p = .04, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

14. Secondary Outcome: The Mean Number of Visits to a Primary Care Provider (PCP) According to Treatment Assignment
Description: At each visit parents were asked if they had taken their child to his/her primary care physician since the last contact. Medical records were also reviewed.
Time Frame: This was assessed at each study visit, i.e. Day 4-5, Day 10-12, Day 21-25, and at interim visits. The last assessment was made at the Day 21-25 visit. The mean day for this latter visit was 22.8.
Population: The analysis was ITT. The participants for analysis were the children with follow-up assessment visits.
Measure: Mean (Standard Deviation); unit: visits to PCP
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 146
visits to PCP | .15 (.40) | .23 (.50)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding visits to primary care provider; Test type: Superiority or Other; p = .20, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

15. Secondary Outcome: The Mean Number of Emergency Room Visits According to Treatment Assignment
Description: At each visit we asked parents if they had to take their child to the emergency department. We also reviewed medical records to assure even more accurate reporting.
Time Frame: as for outcome 14
Population: The analysis was ITT. The participants for analysis were the children with follow-up assessment visits.
Measure: Mean (Standard Deviation); unit: visits to ER
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 146
visits to ER | .07 (.26) | .07 (.25)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding visits to emergency room; Test type: Superiority or Other; p = .90, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

16. Primary Outcome: The Time to Resolution of Symptoms, Defined as Acute Otitis Media-Severity of Symptoms (AOM-SOS) Score of 0 or 1, According to Treatment Assignment
Description: Time to resolution of symptoms is defined as the time from randomization until a child's AOM-SOS score reaches 0 or 1. The parent rated each of 7 symptoms (ear tugging, crying, irritability, difficulty sleeping, diminished activity, diminished appetite & fever) as 0, 1 or 2 (none, a little, a lot) and recorded the ratings in a diary following enrollment on Day 1, twice daily Days 2 and 3, then once daily Days 4-7. Each set of ratings was summed to obtain an AOM-SOS score. The maximum possible score was 14 and the minimum was 0. A score >=3 was required to be enrolled in the study.
Time Frame: The first 7 days on therapy
Population: The analysis was ITT. The number of participants is equal to the number of children randomized.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 144 | 147
participants
  Resolved by Day 1 - PM | 20 | 9
  Censored by Day 1 - PM | 1 | 2
  Resolved by Day 2 - AM | 38 | 28
  Censored by Day 2 - AM | 1 | 2
  Resolved by Day 2 - PM | 50 | 41
  Censored by Day 2 - PM | 1 | 3
  Resolved by Day 3 - AM | 70 | 58
  Censored by Day 3 - AM | 1 | 3
  Resolved by Day 3 - PM | 77 | 66
  Censored by Day 3 - PM | 1 | 4
  Resolved by Day 4 | 87 | 78
  Censored by Day 4 | 1 | 4
  Resolved by Day 5 | 96 | 92
  Censored by Day 5 | 1 | 4
  Resolved by Day 6 | 110 | 98
  Censored by Day 6 | 1 | 4
  Resolved by Day 7 | 114 | 106
  Censored by Day 7 | 30 | 41
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the time to resolution of symptoms where resolution is defined as AOM-SOS score <=1; Test type: Superiority or Other; p = .14, Regression, Cox; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children; Hazard Ratio (HR) = 1.22 — The Amoxicillin-Clavulanate arm represents the numerator and the Placebo arm represents the denominator

17. Primary Outcome: The Time to Resolution of Symptoms, Defined as Acute Otitis Media-Severity of Symptoms (AOM-SOS) Score of 0 or 1 on Two Consecutive Occasions, According to Treatment Assignment
Description: Time to resolution of symptoms is defined as the time from randomization until a child's AOM-SOS score reaches <= 1 on two consecutive occasions. The parent rated each of 7 symptoms (ear tugging, crying, irritability, difficulty sleeping, diminished activity, diminished appetite & fever) as 0, 1 or 2 (none, a little, a lot) & recorded the ratings in a diary following enrollment on Day 1, twice daily Days 2 & 3, & once daily Days 4-7. Each set of ratings was summed to obtain an AOM-SOS score. The maximum possible was 14 and the minimum 0. A score >=3 was required to be enrolled in the study.
Time Frame: The first 7 days on therapy
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 144 | 147
participants
  Resolved by Day 1 - PM | 0 | 0
  Censored by Day 1 - PM | 1 | 2
  Resolved by Day 2 - AM | 17 | 8
  Censored by Day 2 - AM | 1 | 2
  Resolved by Day 2 - PM | 29 | 20
  Censored by Day 2 - PM | 1 | 3
  Resolved by Day 3 - AM | 34 | 29
  Censored by Day 3 - AM | 1 | 3
  Resolved by Day 3 - PM | 50 | 42
  Censored by Day 3 - PM | 1 | 4
  Resolved by Day 4 | 58 | 51
  Censored by Day 4 | 1 | 5
  Resolved by Day 5 | 70 | 63
  Censored by Day 5 | 1 | 5
  Resolved by Day 6 | 80 | 69
  Censored by Day 6 | 1 | 5
  Resolved by Day 7 | 96 | 76
  Censored by Day 7 | 48 | 71
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the time to resolution of symptoms where resolution is defined as AOM-SOS score <=1 on two consecutive occasions; Test type: Superiority or Other; p = .04, Regression, Cox; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children; Hazard Ratio (HR) = 1.37 — The Amoxicillin-Clavulanate arm represents the numerator and the Placebo arm represents the denominator

18. Secondary Outcome: The Mean Number of Antibiotic Prescriptions, Exclusive of Study Medication, According to Treatment Assignment
Description: This is the number of times, in the course of the study, a child required treatment with an antibiotic other than the blinded study medication.
Time Frame: as for outcome 14
Population: The analysis was ITT. The participants for analysis were the children with follow-up.
Measure: Mean (Standard Deviation); unit: antibiotic prescriptions
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 146
antibiotic prescriptions | .35 (.58) | .75 (.73)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the number of antibiotic prescriptions, exclusive of the blinded study medication; Test type: Superiority or Other; p < .001, Generalized estimating equations; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

19. Secondary Outcome: The Total Number of Visits, Summed Across All Participants, at Which a Family Member Reported Having Missed Work According to Treatment Assignment
Description: At each visit, parent or parents were asked if their child's illness had caused either parent to miss a day or partial day of work. The total number of visits is summed across all participants in the respective treatment arms.
Time Frame: as for outcome 14
Population: The analysis was ITT. The participants for analysis were the children with follow-up assessment visits.
Measure: Number; unit: visits
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 146
visits | 33 | 33
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the visits at which family member reported missing work, i.e. number of such visits / total number of follow-up assessment visits; Test type: Superiority or Other; p = .93, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

20. Secondary Outcome: The Total Number of Visits, Summed Across All Participants, at Which a Family Member Reported Making Special Daycare Arrangements According to Treatment Assignment
Description: At each visit, parent or parents were asked if their child's illness had caused them to make alternative daycare arrangements. The total number of visits is summed across all participants in the respective treatment arms.
Time Frame: as for outcome 14
Population: The analysis was ITT. The participants for analysis were the children with follow-up assessment visits.
Measure: Number; unit: visits
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 146
visits | 22 | 24
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two groups regarding the visits at which family member reported making special daycare arrangements, i.e. number of such visits / total number of follow-up assessment visits; Test type: Superiority or Other; p = .66, Generalized estimating equations; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

21. Secondary Outcome: The Mean Score Representing Parental Satisfaction With the Study Medication As Recorded at the On-therapy Visit According to Treatment Assignment
Description: Parents were asked to circle the expression that best represented their satisfaction with the study medication. These expressions have an assigned value: Very dissatisfied = 1, Somewhat dissatisfied = 2, Neither satisfied nor dissatisfied = 3, Somewhat satisfied = 4 and Very satisfied = 5.
Time Frame: On-therapy visit. The mean day for this visit was 5.0.
Population: The analysis was ITT. The number of participants equals the number of children whose parent reported a satisfaction score at the on-therapy visit.
Measure: Mean (Standard Deviation); unit: parental satisfaction score
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 139 | 142
parental satisfaction score | 4.19 (0.97) | 4.13 (1.06)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the groups regarding the mean parental satisfaction score at the on-therapy visit; Test type: Superiority or Other; p = .71, Regression, Linear; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

22. Secondary Outcome: The Mean Score Representing Parental Satisfaction With the Study Medication As Recorded at the End-of-therapy Visit According to Treatment Assignment
Description: as for outcome 21
Time Frame: End-of-therapy visit. The mean day for this visit was 11.6.
Population: The analysis was ITT. The number of participants equals the number of children whose parent reported a satisfaction score at the end-of-therapy visit.
Measure: Mean (Standard Deviation); unit: parental satisfaction score
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 138 | 140
parental satisfaction score | 4.40 (0.92) | 4.12 (1.16)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the groups regarding the mean parental satisfaction score at the end-of-therapy visit; Test type: Superiority or Other; p = .04, Regression, Linear; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

23. Secondary Outcome: The Mean Score Representing Parental Satisfaction With the Study Medication As Recorded at the Follow-up Visit According to Treatment Assignment
Description: as for outcome 21
Time Frame: Follow-up visit. The mean day for this visit was 22.8.
Population: The analysis was ITT. The number of participants equals the number of children whose parent reported a satisfaction score at the follow-up visit.
Measure: Mean (Standard Deviation); unit: parental satisfaction score
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 139 | 139
parental satisfaction score | 4.53 (0.89) | 4.17 (1.12)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the groups regarding the mean parental satisfaction score at the follow-visit visit; Test type: Superiority or Other; p = .005, Regression, Linear; The comparison adjusted for site, history of recurrent acute otitis media and exposure to other children

24. Primary Outcome: The Weighted Average Acute Otitis Media - Severity of Symptom (AOM-SOS) Score, According to Treatment Assignment
Description: The AOM-SOS score is derived from parent scoring each of 7 symptoms (ear tugging, crying, irritability, difficulty sleeping, diminished activity, diminished appetite & fever) associated with AOM as 0, 1 or 2 (none, a little, a lot). The AOM-SOS was administered twice daily the first 3 days of follow-up, then daily for 4 additional days. Symptom burden for each child is determined by calculating the weighted average of symptom scores post-enrollment over the first 7 days of therapy. Scores are weighted by 1/k, where k is the number of post-enrollment assessments taken on that day.
Time Frame: During the first 7 days of therapy
Population: The analysis was ITT. The number of participants equals the number of children with at least one AOM-SOS score post-enrollment in the first 7 days of therapy. The score was based on diaries completed at home by the child's parent.
Measure: Mean (Standard Error); unit: AOM-SOS score
Arm/Group | Amoxicillin-Clavulanate | Placebo
Number analyzed (Participants) | 143 | 144
AOM-SOS score | 2.79 (0.16) | 3.42 (0.18)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate vs Placebo; Null hypothesis: There is no difference between the two treatment groups regarding the mean weighted average acute otitis media - severity of symptom (AOM-SOS) score (symptom burden), post-enrollment, over the first 7 days of therapy; Test type: Superiority or Other; p = .01, Regression, Linear; The comparison was adjusted for site, history of recurrent acute otitis media and exposure to other children

ADVERSE EVENTS:
Time Frame: We monitored children and queried parents regarding adverse events at each study visit, i.e. Day 4-5, Day 10-12, and Day 21-25, and at interim visits. The last assessment was made at the Day 21-25 visit. The mean day for this latter visit was 22.8.
Description: A condition present at enrollment was recorded in the Review of Systems, not as an Adverse Event. However, if this condition worsened or developed after the enrollment visit, we reported this as an Adverse Event.
Arm/Group | Amoxicillin-Clavulanate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/144 | 2/147
Other Adverse Events (participants affected / at risk) | 117/144 | 104/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-Clavulanate (N=144) | Placebo (N=147)
Mastoiditis (Ear and labyrinth disorders) | 0 (0) | 1 (1) — One child was diagnosed with an early mastoiditis at the on-therapy visit. Middle ear culture yielded serotype 19A S. pneumoniae. The child was hospitalized and recovered uneventfully.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — One child developed pneumonia on study day three. The child was hospitalized and recovered uneventfully. After discharge the mother withdrew from the study. She felt it was too burdensome to complete the memory aid and come for follow-up visits.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-Clavulanate (N=144) | Placebo (N=147)
Asthma or wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (10)
Conjunctivitis (Eye disorders) | 6 (6) | 11 (12)
Diaper dermatitis (Skin and subcutaneous tissue disorders) | 80 (91) | 57 (64)
Fever (General disorders) | 8 (8) | 8 (8)
Gastroenteritis (Gastrointestinal disorders) | 7 (7) | 9 (9)
Oral thrush (Gastrointestinal disorders) | 7 (7) | 1 (1)
Protocol defined diarrhea (Gastrointestinal disorders) | 36 (40) | 24 (25) — This is defined as 3 watery stools in 1 day or 2 watery stools for each of 2 consecutive days.
Teething (General disorders) | 12 (13) | 15 (15)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 33 (35) | 34 (36)
Viral exanthem (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Viral illness (General disorders) | 6 (6) | 6 (6)
Vomiting (Gastrointestinal disorders) | 15 (18) | 16 (16)

LIMITATIONS AND CAVEATS:
Long-term implications of abnormal otoscopic findings (bulging) without symptoms, and persistent middle-ear effusion without findings of acute inflammation as forerunners of subsequent acute otitis media episodes remains uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes